CLINICAL TRIAL: NCT03474549
Title: Treatment With Intent to Generate Endovascular Reperfusion
Acronym: TIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-TI-001
Record Dates: First submitted 2018-03-06; First posted 2018-03-22 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke
Keywords: Mechanical thrombectomy,; Brain; Brain clot; Brain infarction; Cerebral ischemia; Neurovascular intervention; Revascularization; Reperfusion; Stent retriever; Tigertriever; Stroke; Rapid Medical
MeSH Terms: conditions — Ischemic Stroke; Brain Infarction; Brain Ischemia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tigertriever revascularization device (Experimental): Mechanical thrombectomy with Tigertriever
  Interventions: Device: Tigertriever revascularization device

INTERVENTIONS:
Device: Tigertriever revascularization device — Mechanical Thrombectomy

SUMMARY:
Tigertriever is a CE marked mechanical revascularization device indicated to restore blood flow by removing thrombus from a large intracranial vessel in patients experiencing ischemic stroke within 8 hours of symptom onset. Patients who are ineligible for IV t-PA or who fail IV t-PA therapy are candidates for treatment.

The objective of the TIGER Study is to evaluate the safety and effectiveness of the Tigertriever device in restoring blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke due to a large vessel occlusion (LVO). This study is designed to support substantial equivalence to approved and marketed products such as the Solitaire or Trevo Retriever.

ELIGIBILITY:
Inclusion Criteria:

1. New focal neurologic deficit consistent with being of acute cerebral ischemia origin.
2. Age 18-85 years old (inclusive).
3. Interventionalist estimates that treatment with the Tigertriever (first deployment in target vessel) can be achieved within 8 hours of symptom onset.
4. Patient either: a) eligible for, and received, IV t-PA within 3 hours of symptom onset, at the correct 0.9 mg/kg dose, or b) ineligible for IV t-PA.
5. NIH Stroke Scale score of 8-29.
6. No known significant pre-stroke disability (prestroke mRS 0 or 1).
7. Catheter angiographic confirmation of a large vessel occlusion in the intracranial internal carotid artery, the M1 or M2 segments of the middle cerebral artery, the intracranial vertebral artery, or the basilar artery that is accessible to Tigertriever device.
8. For strokes in the anterior circulation, the following imaging criteria should also be met:

   1. MRI criterion: volume of diffusion restriction visually assessed ≤50 mL, OR
   2. CT criterion: ASPECTS 6 to 10 on baseline NCCT or CTA-source images,
9. For strokes in the posterior circulation, the following imaging criterion should also be met: pcASPECTS score 8 to 10 on baseline NCCT, CTA-source images, or DWI MRI.
10. Anticipated life expectancy of at least 6 months.
11. A signed informed consent by patient or a Legally Authorized Representative or independent physician in case of oral consent.

Exclusion Criteria:

1. Subject already participating in another study of an investigational treatment device or treatment.
2. Use of any other intra-arterial recanalization drug or device prior to the Tigertriever (Tigertriever not as first choice device).
3. Angiographically evident excessive arterial tortuosity precluding device access to the thrombus.
4. For all patients, severe sustained hypertension with SBP >220 and/or DBP >120; for patients treated with IV tPA, sustained hypertension despite treatment with SBP >185 and/or DBP > 110.
5. Glucose < 50 mg/dl (2.78 mmol/L) or > 400 mg/dl (22.20 mmol/L).
6. Known hemorrhagic diathesis.
7. Coagulation factor deficiency or oral anti-coagulant therapy with an international normalized ratio (INR) of more than 3.0.
8. Treatment with heparin within 48 h with a partial thromboplastin time more than two times the laboratory normal.
9. Patients who have received a direct thrombin inhibitor within the last 48 hours; must have a partial thromboplastin time (PTT) less than 1.5 times the normal to be eligible.
10. Platelet count of less than 50,000/uL.
11. History of severe allergy to contrast medium, nickel, or Nitinol.
12. Intracranial hemorrhage.
13. Significant mass effect with midline shift.
14. Intracranial tumor (apart from small meningioma, ≤ 2 cm in diameter).
15. Stenosis or any occlusion in the deployment site or in a proximal vessel requiring treatment or preventing device access to the thrombus (for example, stenosis or occlusion in the cervical internal carotid artery).
16. Females who are pregnant or breastfeeding.
17. Known current use of cocaine at time of treatment.
18. Prior recent stroke in the past 3 months.
19. Renal failure with serum creatinine >3.0 or Glomerular Filtration Rate (GFR) <30.
20. Known cerebral vasculitis.
21. Rapidly improving neurological status defined as improvement of greater than 8 points on the NIHSS or improvement to NIHSS of < 6 prior to procedure
22. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
23. Ongoing seizure due to stroke.
24. Evidence of active systemic infection.
25. Known cancer with metastases.
26. Suspicion of aortic dissection, septic embolus, or bacterial endocarditis.
27. Evidence of dissection in the extra or intracranial cerebral arteries.
28. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
29. Aneurysm in target vessel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Saver, Dr., Principal Investigator — Geffen School of Medicine at UCLA; Rishi Gupta, Dr., Principal Investigator — WellStar Medical Group
Locations (17):
- United States (16):
  - UCLA medical center, Los Angeles, California
  - Los Robles, Thousand Oaks, California
  - Tenet Health, Coral Springs, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Baptist Health South Florida, Miami, Florida
  - University of Miami, Miami, Florida
  - WellStar Research Institute, Marietta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Massachusetts, Worcester, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - University of Buffalo, Buffalo, New York
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy Health, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - VBMC Harlingen, Harlingen, Texas
- Rambam, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta R, Saver JL, Levy E, Zaidat OO, Yavagal D, Liebeskind DS, Khaldi A, Gross B, Lang M, Narayanan S, Jankowitz B, Snyder K, Siddiqui A, Davies J, Lin E, Hassan A, Hanel R, Aghaebrahim A, Kaushal R, Malek A, Mueller-Kronast N, Starke R, Bozorgchami H, Nesbit G, Horikawa M, Priest R, Liu J, Budzik RF, Pema P, Vora N, Taqi MA, Samaniego E, Wang QT, Nossek E, Dabus G, Linfante I, Puri A, Abergel E, Starkman S, Tateshima S, Jadhav AP; TIGER Trial Investigators. New Class of Radially Adjustable Stentrievers for Acute Ischemic Stroke: Primary Results of the Multicenter TIGER Trial. Stroke. 2021 May;52(5):1534-1544. doi: 10.1161/STROKEAHA.121.034436. Epub 2021 Mar 19. PMID 33739136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tigertriever Revascularization Device
Started | 160
Completed | 123
Not Completed | 37
Not completed — Death | 31
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 160 subjects enrolled
Arm/Group | Tigertriever Revascularization Device
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 134
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Successful Reperfusion, Defined as mTICI Score ≥ 2b
Description: Effectiveness (Successful reperfusion)
Time Frame: Day 0 (end of procedure)
Population: main study cohort (post lead-in)- 117 overall patients (including lead-in)- 160
Measure: Count of Participants; unit: Participants
Arm/Group | Tigertriever Revascularization Device
Number analyzed (Participants) | 160
Participants | 130

2. Primary Outcome: All-cause Mortality
Description: Safety (All-cause mortality)
Time Frame: 90 days post treatment
Population: main study cohort (post lead-in)- 117 all patients (including lead-in)- 160
Measure: Count of Participants; unit: Participants
Arm/Group | Tigertriever Revascularization Device
Number analyzed (Participants) | 160
Participants | 31

3. Primary Outcome: Symptomatic Intracranial Hemorrhage (sICH) Defined as Any Parenchymal Hematoma Type 2, Remote Intracerebral Hemorrhage, Subarachnoid Hemorrhage, or Intraventricular Hemorrhage That is the Predominant Cause of ≥4 Point NIHSS Deterioration at 24 Hours
Description: Safety (Symptomatic intracranial hemorrhage (sICH)) defined as any parenchymal hematoma type 2, remote intracerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage that is the predominant cause of ≥4 point NIHSS deterioration at 24 hours.
Time Frame: 24 hours post procedure
Population: main study cohort (post lead-in)- 117 overall patients (including lead-in)- 160
Measure: Count of Participants; unit: Participants
Arm/Group | Tigertriever Revascularization Device
Number analyzed (Participants) | 160
Participants | 3

4. Secondary Outcome: Modified Rankin Scale (mRS) Score of ≤2
Description: modified Ranking Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
Time Frame: 90 days post treatment
Population: Sample sizes vary due to missing data at 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Tigertriever Revascularization Device
Number analyzed (Participants) | 154
Participants | 86

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Tigertriever Revascularization Device
All-Cause Mortality (participants affected / at risk) | 31/160
Serious Adverse Events (participants affected / at risk) | 71/160
Other Adverse Events (participants affected / at risk) | 120/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigertriever Revascularization Device (N=160)
Cardiac disorders (Cardiac disorders) | 15
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3
Gastrointestinal disorders (Gastrointestinal disorders) | 4
General disorders and administration site conditions (General disorders) | 2
Infections and infestations (Infections and infestations) | 5
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorders|Psychiatric disorders (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders (Nervous system disorders) | 17
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4
Surgical and medical procedures (Surgical and medical procedures) | 1
Vascular disorders (Vascular disorders) | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tigertriever Revascularization Device (N=160)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 16 (16)
Cardiac disorders (Cardiac disorders) | 21 (21)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 18
General disorders and administration site conditions (General disorders) | 5
Infections and infestations (Infections and infestations) | 7
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 5
Investigations (Investigations) | 2
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Nervous system disorders (Nervous system disorders) | 18
Renal and urinary disorders (Renal and urinary disorders) | 3
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures (Surgical and medical procedures) | 1
Vascular disorders (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03474549/Prot_SAP_000.pdf